CLINICAL TRIAL: NCT01111916
Title: A Development Study Using Vaginal Tactile Imager to Assess the Elasticity Properties of the Vaginal Wall and Surrounding Connective Tissue
Brief Title: Development Study Using Vaginal Tactile Imager
Status: Completed | Type: Observational
Sponsor: Artann Laboratories (Industry)
Collaborators: National Institute on Aging (NIA) (NIH); Princeton Healthcare System (Other)
Responsible Party: Sponsor
Other Study IDs: VTI 02; 1R43AG034714-01 (NIH)
Record Dates: First submitted 2010-03-22; First posted 2010-04-28 (Estimated); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective is to evaluate and optimize tactile imaging technology in evaluation of tissue elasticity parameters in the female pelvis.

DETAILED DESCRIPTION:
Pelvic organ prolapse affects 40-50% of women in US. This study aims to establish a reliable examination procedure, collect data necessary for assessing the performance of Vaginal Tactile Imaging sensors, assess clinical suitability of interface software and correlate elasticity measurements with clinical examination findings for normal versus prolapse conditions of the female pelvis.

ELIGIBILITY:
Inclusion Criteria:

1. no evidence of pelvic organ prolapse and no prior pelvic surgery
2. stage 1 or greater pelvic organ prolapse affecting one or more vaginal compartments
3. no evidence of pelvic organ prolapse with prior pelvic surgery (with or without the use of graft material)

Exclusion Criteria:

1. patients with active skin infection, tissue breakdown or ulceration
2. patients with abnormal vaginal anatomy, including vaginal septum, history of vaginal/pelvic radiation, presence of a vaginal tumor or lesion
3. recent pelvic surgery with less than 3-month interval from surgery

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult women with normal pelvic anatomy
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2010-03; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
To determine whether there is a detectable difference in 3-D elasticity images provided by Vaginal Tactile Imager for the patients with presence or absence of prolapse. | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Egorov, PhD, Principal Investigator — Artann Laboratories
Locations (2):
- United States (2):
  - Princeton Urogynecology, Princeton, New Jersey
  - Institute for Female Pelvic Medicine and Reconstructuve Surgery, Allentown, Pennsylvania

REFERENCES:
- [Result] Egorov V, van Raalte H, Lucente V. Quantifying vaginal tissue elasticity under normal and prolapse conditions by tactile imaging. Int Urogynecol J. 2012 Apr;23(4):459-66. doi: 10.1007/s00192-011-1592-z. Epub 2011 Nov 10. PMID 22072417
- [Result] Egorov V, Patel M, Sarvazyan AP. Vaginal tactile imager for direct tissue elasticity modulus estimation. Proceedings of the 10th International Tissue Elasticity Conference, Arlington, Texas, October 12-15, 2011:59.
- [Result] Egorov V, van Raalte H, Lucente V. Vaginal tactile imaging: clinical results. Proceedings of the 10th International Tissue Elasticity Conference, Arlington, Texas, Oct 12-15, 2011: 66.
- [Result] van Raalte H, Lucente V, Egorov V. 3-D imaging and quantifying vaginal tissue elasticity under normal and prolapse conditions. International Urogynecological Association: 36th Annual Meeting, Lisbon, Portugal, June 28 - July 2, 2011.
- [Result] van Raalte H, Egorov V, Lucente V. Tactile imaging of pelvic floor changes with age and parity. American Urogynecologic Society: 32nd Annual Scientific Meeting, Providence, Rhode Island, September 14-17, 2011.